CLINICAL TRIAL: NCT01530477
Title: DXA Precision and Accuracy Comparison Study
Acronym: DXA P&A
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination due to inability to meet enrollment for >350lb weight class
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 101.02-2011-GES-0005
Record Dates: First submitted 2012-02-06; First posted 2012-02-10 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-08

CONDITIONS: Osteopenia
Keywords: Bone mineral density; weight; body composition; DEXA; DXA
MeSH Terms: conditions — Bone Diseases, Metabolic; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Skeletal (Experimental): Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of three systems [Lunar Prodigy (GEHC), Lunar iDXA (GEHC) and Discovery A (Hologic)], and 60 will be measured on all three systems [Lunar Prodigy (GEHC), Lunar iDXA (GEHC) and Discovery A (Hologic)],(total of evaluable 90 subjects).
  ** Subjects can enroll in both Skeletal and Body Composition cohorts. Analysis will be performed within each cohort.**
  Interventions: Device: Lunar Prodigy (GEHC); Device: Lunar iDXA (GEHC); Device: Discovery A (Hologic
- Body Composition (Experimental): Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of the three systems [Lunar Prodigy (GEHC), Lunar iDXA (GEHC) and Discovery A (Hologic)], and 60 will be measured on all three systems [Lunar Prodigy (GEHC), Lunar iDXA (GEHC) and Discovery A (Hologic)], (total of evaluable 90 subjects).
  ** Subjects can enroll in both Skeletal and Body Composition cohorts. Analysis will be performed within each cohort.**
  Interventions: Device: Lunar Prodigy (GEHC); Device: Lunar iDXA (GEHC); Device: Discovery A (Hologic
- Skeletal & Body Composition (Experimental): "Skeletal and Body Composition" was not a cohort that was actively recruited to, it is a cohort for reporting purposes. Subjects will be measured on two of three systems [Lunar Prodigy (GEHC), Lunar iDXA (GEHC) and Discovery A (Hologic)]Subjects were able to consent and enroll to both Skeletal and Body Composition cohorts and these subjects will be counted for under this joint cohort.
  Interventions: Device: Lunar Prodigy (GEHC); Device: Lunar iDXA (GEHC); Device: Discovery A (Hologic

INTERVENTIONS:
Device: Lunar Prodigy (GEHC) — Lunar Prodigy (GEHC) used to obtain Skeletal, and/or Body Composition measurements
Device: Lunar iDXA (GEHC) — Lunar iDXA (GEHC) used to obtain Skeletal, and/or Body Composition measurements
Device: Discovery A (Hologic — Discovery A (Hologic) used to obtain Skeletal, and/or Body Composition measurements

SUMMARY:
This study is being conducted to examine the performance of three common DXA machines (1) Lunar iDXA, (2) Lunar Prodigy and (3) Hologic Discovery A in measuring bone density and body fat.

DETAILED DESCRIPTION:
For this study, two specific groups of volunteers will be recruited. In one group, the scan will measure bone density and in the other group the scan will measure fat. The groups will be broken into weight groups to determine which of the scanners the subject will be scanned on. Subjects will have the option to participate in either one or both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women > 20 years old
2. Willing to provide consent
3. Falls into one of three weight categories, with minimum 30 subjects per category.

   * Less than 200 lbs.
   * 200 (inclusive) to less than 350 lbs.
   * 350 (inclusive) to less than 450 lbs.
4. Participate in only one weight category in either skeletal or body composition cohort, or both.

Exclusion Criteria:

1. Inability to remain still for the duration of the DXA scans as judged by study Investigator.
2. Un-removable internal / external scan artifacts e.g. plaster casts, metal rodding naso-gastric tubes, etc.
3. Females of childbearing potential* with actual (confirmed by positive urine pregnancy test) or suspected (based on study Investigator evaluation despite a negative urine test) pregnancy.
4. Subject had already given consent to participate in any aspect of this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Miller, MD, Principal Investigator — Study site
Locations (1):
- Colorado Center for Bone Research, Lakewood, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 subjects consented for the Skeletal Cohort only. A total of 12 subjects consented for the Body Composition Cohort only. A total of 53 subjects consented to participate in both the Skeletal and Body Composition cohorts. Recruitment occurred at the primary site from January to December 2012.
Pre-assignment Details: Subjects were able to consent and participate in one or both cohorts (Outcome Measure Reporting Groups: Skeletal and Body Composition). GE prematurely ended the study with 82 consented individuals but a total of 135 scans were acquired across the cohorts.
Groups:
- Skeletal: Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of the three systems, and 60 will be measured on all three systems (total of evaluable 90 subjects). Subjects willing to participate in Skeletal & Body Composition are counted towards the 90 evaluable subject requirement of the protocol for the Skeletal Cohort.
- Body Composition Only: Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of the three systems, and 60 will be measured on all three systems (total of evaluable 90 subjects). Subjects willing to participate in Skeletal & Body Composition are counted towards the 90 evaluable subject requirement of the protocol for the Body Composition Cohort.
- Skeletal & Body Composition: "Skeletal & Body Composition" was not a cohort that was actively recruited to, it is a cohort for reporting purposes. Subjects were able to consent and enroll to both Skeletal and Body Composition cohorts and these subjects will be counted for under this joint cohort.
Period: Overall Study
Arm/Group | Skeletal | Body Composition Only | Skeletal & Body Composition
Started | 17 (17 subjects consented to the Skeletal cohort only.) | 12 (12 subjects consented to the Body Composition cohort only.) | 53 (53 subjects consented to both the Skeletal and body Composition cohorts.)
Completed | 17 (17 subjects completed imaging in the Skeletal cohort only.) | 12 (12 subjects completed imaging in the Body Composition cohort only.) | 53 (53 subjects completed the imaging in both the Skeletal and Body Composition cohorts.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Body Composition: Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of the three systems, and 60 will be measured on all three systems (total of evaluable 90 subjects). Subjects willing to participate in Skeletal & Body Composition are counted towards the 90 evaluable subject requirement of the protocol for the Body Composition Cohort.
- Skeletal and Body Composition: "Skeletal and Body Composition" was not a cohort that was actively recruited to, it is a cohort for reporting purposes. Subjects were able to consent and enroll to both Skeletal and Body Composition cohorts and these subjects will be counted for under this joint cohort.
- Total: Total of all reporting groups
Arm/Group | Skeletal | Body Composition | Skeletal and Body Composition | Total
Number analyzed (Participants) | 17 | 12 | 53 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 12 | 53 | 82
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 25 | 39
  Male | 9 | 6 | 28 | 43

OUTCOME MEASURES:

1. Primary Outcome: Short Term Precision Comparison Across Three DXA Devices
Description: BMD precision will be reported across three DXA devices in major skeletal and body composition sites. The short-term precision was calculated as RMS-SD (root mean square standard deviation) over the mean for each cohort. The skeletal cohort will not have short-term precision value for body composition indexes due to the different region of measurement. The same will apply to the body composition cohort. As the result, the "Skeletal & Body Composition" cohort identified in participant flow and overall study summary will not have an analysis provided.
Time Frame: Less than 6 months
Measure: Number; unit: Percentage of variance
Arm/Group | Skeletal | Body Composition Only
Number analyzed (Participants) | 70 | 65
Percentage of variance
  iDXA Spine BMD | 1.0 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Prodigy Spine BMD | 1.3 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Discovery A Spine BMD | 1.2 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  iDXA Femural neck BMD | 1.5 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Prodigy Femural neck BMD | 1.6 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Discovery A Femural neck BMD | 2.1 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  iDXA Total Femur BMD | 0.8 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Prodigy Total Femur BMD | 0.8 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  Discovery A Total Femur BMD | 0.7 | NA — This "Skeletal" region of interest is not available in the "Body Composition" cohort.
  iDXA Total Body BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 0.8
  Prodigy Total Body BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 0.9
  Discovery A Total Body BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 1.9
  IDXA Trunk BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 1.0
  Prodigy Trunk BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 1.2
  Discovery A Trunk BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 5.8
  iDXA Leg BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 0.8
  Prodigy Leg BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 1.3
  Discovery A Leg BMD | NA — This "Body Composition" cohort region of interest is not available in the "Skeletal" cohort. | 1.9

ADVERSE EVENTS:
Groups:
- Skeletal; Body Composition: Recruitment for each cohort will include approximately equal male/female split (no gender bias). Depending on the weight category, for each cohort, a minimum of 30 adult subjects will be measured on two of the three systems, and 60 will be measured on all three systems (total of evaluable 90 subjects).
Arm/Group | Skeletal | Body Composition
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/65
Other Adverse Events (participants affected / at risk) | 0/70 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less